CLINICAL TRIAL: NCT05537753
Title: Encore PFO Closure Device U.S. IDE Randomized Trial - The PerFOrm Trial
Brief Title: Encore PFO Closure Device - The PerFOrm Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Encore Medical Inc. (Industry)
Collaborators: Bright Research Partners (Industry); Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENC-CL-5000
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Patent Foramen Ovale; Cryptogenic Stroke
Keywords: PFO closure; Stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Encore PFO closure device (Experimental)
  Interventions: Device: Encore PFO closure device
- Any FDA-approved PFO closure device chosen by the investigator (Active Comparator)
  Interventions: Device: FDA-approved PFO closure device

INTERVENTIONS:
Device: Encore PFO closure device — The Encore PFO closure device comprises an implant component and a single-use delivery system.
  Arms: Encore PFO closure device
Device: FDA-approved PFO closure device — Chosen by the investigator
  Arms: Any FDA-approved PFO closure device chosen by the investigator

SUMMARY:
The objective of this study is to establish reasonable assurance of safety, effectiveness, and noninferiority of the Encore PFO closure device when compared to any investigator chosen FDA-approved PFO closure device.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized clinical study to determine the safety and effectiveness of the Encore PFO closure device, which is indicated for percutaneous, transcatheter closure of a patent foramen ovale (PFO) in patients who have had a cryptogenic stroke due to a presumed paradoxical embolism.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PFO, defined as visualization of microbubbles per TEE in the left atrium within three cardiac cycles from the right atrial opacification demonstrating right-to-left shunting at rest and/or during Valsalva release
2. Cryptogenic stroke within the last 270 days; stroke is defined as acute focal neurological deficit, presumed to be due to focal ischemia, and confirmed by MRI or CT to be a new, neuroanatomically relevant cerebral infarct

Exclusion Criteria:

1. Age <18 years and age >60 years
2. Greater than 50% lumen diameter stenosis of intracranial or extracranial vessels
3. Intracardiac thrombus or tumor
4. Acute or recent (within 6 months) myocardial infarction (MI) or unstable angina
5. Left ventricular aneurysm or akinesis
6. Mitral valve stenosis (mitral valve area less than 1.5cm2) or severe mitral regurgitation
7. Aortic valve stenosis (gradient >40 mmHg) or severe aortic valve regurgitation
8. Mitral or aortic valve vegetation or prosthesis
9. Left ventricular ejection fraction <35%
10. Other identifiable cause of stroke, including but not limited to aortic arch plaques (protruding >4 mm into the lumen), large artery atherosclerotic disease, an established cardioembolic source, small-vessel occlusive disease, or arterial dissection
11. Evidence of a hypercoagulable disorder requiring anticoagulation therapy; this determination will be based on the evaluation of: anticardiolipin antibody (Ab) of the IgG or IgM type, Lupus anticoagulant, B2-glycoprotein-1 Ab, and fasting plasma homocysteine
12. Another source of right-to-left shunts identified at baseline, including an atrial septal defect and/or fenestrated septum
13. Any history of atrial fibrillation/atrial flutter (chronic or intermittent)
14. Active endocarditis or other untreated infections
15. Chronic kidney disease stage 4 or higher or end-stage renal failure requiring dialysis (eGFR less than 30)
16. Severe liver disease (ALT 3X ULN) or documented cirrhosis
17. Lung disease requiring continuous home oxygen
18. Uncontrolled hypertension, defined as sustained elevated blood pressure >160/90 mm Hg on medication
19. Uncontrolled diabetes mellitus, defined as HbA1c greater than 9 (based on most recent test which must have been collected within the last year)
20. Anatomical or physiological structures that do not permit TEE
21. Anticipated need for treatment of structural cardiac defects other than PFO
22. Concomitant cardiac anomalies requiring an operative procedure
23. Hemorrhagic diseases (e.g., coagulopathy, tendency to hemolysis)
24. Hypersensitivity to contrast medium or nickel
25. Contraindication to aspirin or clopidogrel
26. The required sheaths cannot be passed through the relevant vessels for access to the PFO
27. Vulnerable patient (e.g., incarcerated or cognitively challenged adults); see Section 7.2.1
28. Subject is unable or unwilling to provide informed consent
29. Subject is unable to comply with the protocol
30. Any other clinical reasons for which the patient would not be an appropriate candidate for the study, as determined by the site investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Safety: The incidence of device- or procedure-related serious adverse events (SAEs) | 6 months
Effectiveness: Effective closure | 6 months
  Defined as shunt grade 0 or I while at rest and during Valsalva as assessed by transesophageal echocardiography (TEE) and bubble study as adjudicated by the echocardiographic core laboratory

SECONDARY OUTCOMES:
Complete closure | 6 months
  Defined as shunt grade 0 while at rest and during Valsalva as assessed by TEE and bubble study as adjudicated by the echocardiographic core laboratory
Occurrence of recurrent symptomatic cryptogenic non-fatal stroke or cardiovascular death | 5 years
Occurrence of transient ischemic attacks (TIA) | 5 years
Occurrence of clinically significant new atrial arrhythmia (including atrial fibrillation) | 5 years
Occurrence of technical success | Procedural
Occurrence of procedural success | Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Nielsen, MD, Principal Investigator — Medical University of South Carolina
Locations (8):
- United States (8):
  - Arkansas Cardiology, Little Rock, Arkansas
  - Southern CA Permanente Medical Group - Kaiser San Diego and Scripps Memorial Hospital, La Jolla, California
  - University of South Florida, Tampa, Florida
  - Mercy One Iowa Heart Center, West Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Jackson Heart Clinic, Jackson, Mississippi
  - CHI Health, Omaha, Nebraska
  - Medical University of South Carolina Gazes Research Institute, Charleston, South Carolina